CLINICAL TRIAL: NCT04616443
Title: Phase Ib Study of the Combination Use of Recombinant Human GM-CSF Type II Herpes Simplex Virus (OH2) Injection (Vero Cells) and HX008 Injection in the Treatment of Melanoma
Brief Title: OH2 Injection in Combination With HX008 for Melanoma.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OH2-I-ST-03
Record Dates: First submitted 2020-08-31; First posted 2020-11-05 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Melanoma
Keywords: Oncolytic Virus
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): The HX008 injection is combined with OH2 injections at 10ˆ6 and 10ˆ7 CCID50/mL at a fixed dose of 200 mg, respectively.
  OH2 will be injected individually in the first week, followed by every two weeks while HX008 will be injected every three weeks after the first injection which will be in the second week.
  Interventions: Biological: OH2 injection; Biological: HX008 injection

INTERVENTIONS:
Biological: OH2 injection — Oncolytic Type 2 Herpes Simplex Virus
Biological: HX008 injection — Recombinant humanized anti-PD-1 monoclonal antibody of injection

SUMMARY:
This phase Ib study evaluates the safety and efficacy of OH2 in combination with HX008, an anti-PD-1 antibody, in patients with Melanoma.

OH2 is an oncolytic virus developed upon genetic modifications of the herpes simplex virus type 2 strain HG52, allowing the virus to selectively replicate in tumors. Meanwhile, the delivery of the gene encoding human granulocyte macrophage colony-stimulating factor (GM-CSF) may induce a more potent antitumor immune response.

DETAILED DESCRIPTION:
The trial is a phase Ib study evaluating the safety and efficacy of OH2 injection combined with HX008 injection in patients with Melanoma.

In the Phase Ib dose escalation trial, two doses (1x10e6, 1x10e7 CCID50/mL) of OH2 will be combined with HX008(at a fixed dose of 200mg) will be tested.

In the Phase Ib dose expansion trial, OH2(1x10e7 CCID50/mL) will be injected individually in the first week, followed by every two weeks while HX008(200 mg) will be injected every three weeks after the first injection which will be in the second week.

Blood samples will be collected and radiological imaging will be performed to evaluate safety and efficacy during the trial. Besides, patients will be subjected to cutaneous swabs, and blood/urine/feces sampling to determine virus shedding. Participating patients will be evaluated for objective response rate, progression free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. The non-operative stage III or stage IV malignant tumor patients with clear diagnosis by pathology.
2. Patients who have failed in conventional treatment (including PD-1 monotherapy) (disease progression or intolerance) or who have failed in previously assisted PD-1 monotherapy (last assisted PD-1 treatment relapse or metastasis within 6 months).
3. Patients with Eastern Collaborative Oncology Group (ECOG) Performance Status ≤ 1, expected survival time more than 3 months.
4. Prior anti-tumor treatment (including endocrine, chemical/ radiotherapy,targeted therapy) was over 4 weeks (more than 6 weeks of discontinuation using nitroso-and mitomycin-based chemotherapy) and was recovered to grade 1 from the side effects of prior treatment.
5. There is at least one measurable lesion that is suitable for intratumoral injection. The measured tumor focus is defined as the longest diameter ≥ 5 mm.
6. Asymptomatic central nervous system metastasis, or treated asymptomatic brain metastasis patients, must be examined by a computerized fault scan (CT) or MRI for disease-free progression, stable for at least 3 months, and at least 4 weeks without steroid medication.
7. (a) WBC≥3.0×109／L，ANC≥2.0×109／L ，PLT≥100×109／L，Hb≥90 g/L； (b) BUN and Scr. were in the upper limit of 1.5 times of the normal value; (c) TBIL≤ 1.5 times the upper limit of the normal value. (d) ALT and AST ≤ 2.5 times the upper limit of normal value; The value of patients with liver metastasis did not exceed 5 times the upper limit of normal value. (e) Coagulation function is normal (PT and APPT are within 1.5 times of the upper limit of normal value).
8. Female subjects and their spouses received effective contraceptives during and within 3 months of treatment.
9. Subjects with herpes in the reproductive organs needed three months after the end of herpes.
10. The informed consent was voluntarily signed and the expected compliance was good.

Exclusion Criteria:

1. Severe medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, severe infection, active digestive tract ulcer, abnormal immune function (including, but not limited to, rheumatoid arthritis, lupus erythematosus, Sjogren's syndrome, etc.).
2. Significant surgery is expected to be performed during the 28-day screening period during the study period.
3. Patients had active infections or unexplained fevers (over 38.5℃)during screening and before the first drug use.
4. Past or present immunodeficiency diseases.
5. The lesions do not meet the requirements of injection capacity(1ml) in the tumor body.
6. Pregnant or lactating women.
7. Other experimental therapies or antiviral therapy are used or are being used within 4 weeks of treatment.
8. Allergy to herpes virus and drug ingredients.
9. History of primary grape-film melanoma or other malignant tumors in the 5 years prior to treatment.
10. History of tuberculosis, or have tuberculosis at the time of screening.
11. Suffering from sudden lung disease, intersex lung disease, intersex pneumonia, pulmonary fibrosis, acute lung disease, radioactive pneumonia etc.
12. Patients with active autoimmune diseases or with a history of autoimmune diseases that may relapse, except for:

    1. Type I diabetes with stable condition after taking a fixed dose of insulin;
    2. Hypothyroidism;
    3. Controlled celiac disease;
    4. Skin diseases that do not require systemic treatment;
    5. Any other disease that does not re-occur without external triggers.
13. Concurrent medical condition requiring the use of cortisol (>10mg/day prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment, except for inhalation or topical corticosteroids no more than 10 mg/day prednisone or equivalent.
14. The researchers believe that there is any reason why the patient is not suitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of dose-limiting toxicity (DLT) of OH2 injection in combination with HX008 injection in patients with melanoma | 21 days after treatment
  According to the version 5.0 of the National Cancer Institute Common Terminology Criteria for Adverse Events, the adverse events during the entire study period are evaluated to observe the dose-limiting toxicity.

SECONDARY OUTCOMES:
The response rate of patients with melanoma receiving OH2 injection in combination with HX008 injection | 18 months
  Tumor evaluation is performed according to RECIST1.1 and iRECIST1.1.
The immunoreactivity of OH2 injection and HX008 injection. | 18 months
  Detection of increased systemic immune Response markers in peripheral blood mononuclear cells by flow cytometer.Detection of complement C3, C4 titer.
The immunogenicity of OH2 injection and HX008 injection. | 18 months
  The immunogenicity of OH2 is evaluated by detection of anti-HSV2 antibodies and anti-GM-CSF antibodies in the blood.The immunogenicity of HX008 is evaluated by detection of anti-PD-1 antibodies in blood by ADA.
The biodistribution and biologic effect of OH2 injection. | 18 months
  The biodistribution of OH2 injection as determined by the concentration of OH2 in blood, urine and feces of participating patients.The biologic effect of OH2 injection as determined by the GM-CSF RNA quantification in fine needle aspiration(FNA) of patients.Expression of GM-CSF in FNA.The original result unit is copies/ul.
The pharmacygenic dynamics (PK) characteristics of HX008 injections in the case of HX008 injections combined with OH2 injections. | 18 months
  Cmax.
Explore the changes in peripheral blood and tumor tissue immune-related indicators during treatment. | 18 months
  Peripheral blood T lymphocyte subtype.The ratio of CD4/CD8 in blood lymphocytes. PD-L1 expression in tumor tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China